CLINICAL TRIAL: NCT04281082
Title: Genetic Polymorphisms of ABCB11 and ABCB4 in Women With Intrahepatic Cholestasis of Pregnancy (ICP) and in Their First Degree Relatives
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, SPYRIDON MICHOPOULOS, Head Of The Gastroenterology Departement, Alexandra Hospital, Athens, Greece
Other Study IDs: AlexandraH ICP
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Cholestasis of Pregnancy
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICP: To study the genetic polymorphisms in pregnant women with ICP and in their first degree relatives
  Interventions: Drug: ursofalk

INTERVENTIONS:
Drug: ursofalk — To study the genetic polymorphisms in pregnant women with ICP treated with ursoflak and in their first degree relatives

SUMMARY:
To assess the occurrence of 11 SNP's in ABCB11 and ABCB4 genes in Greek women with ICP compared with healthy pregnant women. Moreover, these genetic polymorphisms will be examined in their first-degree relatives.

DETAILED DESCRIPTION:
Introduction: ICP is commolnly manifested in the 2nd and especially in the 3rd trimester of pregnancy. Pathogenesis of ICP is multifactorial implicating genetic, environmental and hormonologic factors. Prevalence of ICP varies. In certain populations in latin America occurrence of ICP is up to 15% of pregnancies. In Caucasian populations incidence of ICP is approximately 1% of pregnancies. Data for the Greek population are scarce. Genes ABCB4 and ABCB11 that are encoding transport proteins in the hepatocyte are implicated in the pathogenesis of ICP.

Aim of the Study: To study the genetic polymorphisms in pregnant women with ICP and in their first degree relatives Patients and Methods: To recruit 100 women with ICP. Analyze the occurrence of 11 SNP's in ABCB11 and ABCB4 genes in women with ICP. As control group will be used pregnant women without ICP or known hepatic disease. In these women the same analysis for SNP's as in women with ICP will be performed. Exclusion criteria: women with known hepatic disease ( HBV, HCV, HIV, HEV, Autoimmune Hepatitis, Drug induced liver injury, cirrhosis) and women with pregnancy related liver disease (pre-eclampsia, acute fatty liver of pregnancy or HELLP syndrome) Inclusion criteria: pregnant women with ICP. Detailed report of medical history, laboratory and clinical data regarding women and the pregnancy. Follow up of laboratory values before and after the begging of treatment with UDCA.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with ICP

Exclusion Criteria:

* women with known hepatic disease ( HBV, HCV, HIV, HEV, Autoimmune Hepatitis, Drug induced liver injury, cirrhosis)
* women with pregnancy related liver disease (pre-eclampsia, acute fatty liver of pregnancy or HELLP syndrome)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women with ICP. Detailed report of medical history, laboratory and clinical data regarding women and the pregnancy. Follow up of laboratory values before and after the begging of treatment with UDCA.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
genetic polymorphisms in pregnant women with ICP and in their first degree relatives | 01/01/2018-31/01/2021

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided